CLINICAL TRIAL: NCT06000124
Title: The Effect of Plyometric Training on the Balance Ability of the Lower Limbs in the Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Collaborators: National Science and Technology Council (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N202207073
Record Dates: First submitted 2023-05-28; First posted 2023-08-21 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2022-08

CONDITIONS: Plyometric Exercise; Elderly; Balance
MeSH Terms: interventions — Plyometric Exercise

STUDY DESIGN:
Intervention Model Description: The experimental group underwent plyometric training three times a week, performing three rounds each session, for a total intervention period of 10 weeks. The control group, on the other hand, engaged in regular exercises during the same intervention period. Before and after the training program, both groups underwent assessments to evaluate their balance abilities, which included the 30-second sit-to-stand test, time up and go test (TUG), functional reach test (FRT), and lower extremity explosiveness test.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: All subjects were randomly assigned to either the control or experimental group to receive their respective exercise programs. The outcomes assessor was blinded to the group allocation of each participant during baseline and post-intervention assessments. No group assignment information was provided to the care providers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plyometric exercises training (Experimental): High knee lifts, squat jumps, lunge cross jumps, squat jumping lunges, and squat jump twists are examples of plyometric exercises suitable for older adults.
  Interventions: Other: Plyometric exercises
- Regulation exercises program (Active Comparator): The regulated exercise program includes the use of elastic bands, Qigong, and dance et al.
  Interventions: Other: Regulation Exercises Program

INTERVENTIONS:
Other: Plyometric exercises — High knee lifts, squat jumps, lunge cross jumps, squat jumping lunges, and squat jump twists are examples of plyometric exercises suitable for older adults.
  Arms: Plyometric exercises training
Other: Regulation Exercises Program — The regulated exercise program includes the use of elastic bands, Qigong, and dance et al.
  Arms: Regulation exercises program

SUMMARY:
For the elderly using plyometric training, there are very few studies on strengthening the explosive power of the lower limbs of the elderly. For example, past studies have explored the effect of high-speed and low-speed plyometric training on the improvement of muscle contraction speed in the elderly over 60 years old. From the past researches, the study found that compared with low-speed training, High-speed training can not only improve muscle strength, but also effectively increase muscle speed and improve life functions. However, studies using plyometric training to improve lower body balance in older adults are scarce and the evidence is scant. Therefore, the purpose of this study is to explore the clinical benefits of plyometric training for improving the balance ability of the lower limbs in the elderly.

DETAILED DESCRIPTION:
Plyometric training is an exercise method that has gained significant popularity in recent years for effectively enhancing explosive power in the lower limbs. It involves rapid and forceful muscle contractions following a quick stretch. This type of training enables the body to generate maximum muscle strength for short durations during exercise. As individuals age, their ability to produce explosive power decreases, particularly in the lower limbs. This decline in explosive power can result in reduced responsiveness to sudden balance disturbances, leading to falls among the elderly and greatly impacting their daily activities. Hence, the objective of this study was to investigate the effects of a 10-week plyometric training program on the balance ability of the lower limbs in elderly individuals.

A total of 38 elderly participants, aged between 65 and 89 years, were randomly assigned to either the experimental group (N=19) or the control group (N=19). The experimental group underwent plyometric training three times a week, performing three rounds each session, for a total intervention period of 10 weeks. The control group, on the other hand, engaged in regular exercises during the same intervention period. Before and after the training program, both groups underwent assessments to evaluate their balance abilities, which included the 30-second sit-to-stand test, time up and go test (TUG), functional reach test (FRT), and lower extremity explosiveness test. To analyze the data, SPSS 18.0 statistical software was used. Independent sample t-tests were employed to compare the baseline values between the two groups and to determine the differences in the 30-second sit-to-stand test, TUG, FRT, and force plate maximum reaction force values after the intervention. Paired samples t-tests were conducted to assess changes in balance performance from pre-test to post-test. The statistical significance level (α) was set at 0.05.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy elderly individuals aged 65 to 89 years, including both healthy older adults and pre-frail individuals.
2. Able to perform activities of daily living independently at home and in the community

Exclusion Criteria:

1. Severe neurological and musculoskeletal disorders of the lower limbs
2. Severe cardiovascular disease
3. Vestibular deficit
4. Medication affects or improves balance ability

Ages: 65 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 38 (Actual)
Dates: Start 2023-02-14 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
30-second sit-to-stand test | From enrollment to the end of treatment at 10 weeks
  1 Instruct the patient: (1) Sit in the middle of the chair. (2) Place your hands on the opposite shoulder crossed, at the wrists. (3) Keep your feet flat on the floor. (4) Keep your back straight, and keep your arms against your chest. (5) On "Go," rise to a full standing position, then sit back down again. (6) Repeat this for 30 seconds. 2 On the word "Go," begin timing. If the patient must use his/her arms to stand, stop the test. Record "0" for the number and score. 3 Count the number of times the patient comes to a full standing position in 30 seconds. If the patient is over halfway to a standing position when 30 seconds have elapsed, count it as a stand. 4 Record the number of times the patient stands in 30 seconds.
time up and go test (TUG) | From enrollment to the end of treatment at 10 weeks
  Patients wear their regular footwear and can use a walking aid, if needed. Begin by having the patient sit back in a standard arm chair and identify a line 3 meters, or 10 feet away, on the floor. 1 Instruct the patient:When I say "Go," I want you to: (1). Stand up from the chair. (2). Walk to the line on the floor at your normal pace. (3). Turn. (4). Walk back to the chair at your normal pace. (5). Sit down again.2 On the word "Go," begin timing. 3 Stop timing after patient sits back down. 4 Record time.
functional reach test (FRT) | From enrollment to the end of treatment at 10 weeks
  Ascertaining dynamic balance.In standing, measures the distance between the length of an outstretched arm in a maximal forward reach, while maintaining a fixed base of support. This information is correlated with risk of falling.

SECONDARY OUTCOMES:
lower extremity explosiveness test | From enrollment to the end of treatment at 10 weeks
  Using force plate to analysis the muscle power in lower extremities.

CONTACTS AND LOCATIONS:
Overall Officials: Chueh-Ho Lin, PhD, Principal Investigator — Taipei Medical University
Locations (1):
- Jiuzhuang Community Development Association, Taipei, Nangang, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD will be shared with other researchers upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: starting in August 2023
Access Criteria: The datasets generated in this study are available from the corresponding author upon reasonable request. PO-CHENG,CHIANG will be review requests.